CLINICAL TRIAL: NCT04011553
Title: The Effectiveness of Virtual Reality Based Rehabilitation in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, EMEL METE, RESEARCH ASSISTANT, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Istanbul Medeniyet University
Record Dates: First submitted 2019-06-24; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Virtual reality; Rehabilitation; Balance; Kinesiophobia
MeSH Terms: conditions — Osteoarthritis, Knee; Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual group (Experimental): This virtual realtiy was implemented with MarVAJED® (Marmara Visual Auditory Joint Education Device) system which was developed by Marmara University, Department of Physiotherapy and Rehabilitation, Istanbul,Turkey. MarVAJED® is a system that evaulates the range of motion of the joints, analyzes the sensation of joint position, provides biofeedback support to increase joint control and the same time allows exercises to be controlled. This device analyzes the joint motion with the help of small sensors (Figure 2). The obtained data transfers to your mobile phone, to the tablet or to your personal computer. It stores the data by downloading it to the central server via internet for storage.
  Interventions: Other: Virtual Reality based Rehabilitation Program
- Control group (Active Comparator): Conventional physiotherapy consists of electrotherapy and exercise programs. Hotpack or coldpack, therapeutic ultrasound (US) and conventional TENS were applied as electrotherapy program.
  Interventions: Other: Virtual Reality based Rehabilitation Program

INTERVENTIONS:
Other: Virtual Reality based Rehabilitation Program — Virtual reality-based rehabilitation was implemented via MarVAJED system. At first the sensors of MarVAJED® were placed under and above the knee joint and then it was calibrated. The content of the game programs included in the MarVAJED system and how to perform these games with the exercises were explained to the participants. We used games called "Crazy Wings and Blasting Ball" included in the MarVAJED®.There was a bird figure in Crazy Wings game and represented knee joint of participants. Although the bird figure moved upwards during knee flexion, it moved downward in knee extension, there were some obstacles on the way of the bird went. The subjects were asked to follow the bird figure visually and to pass through the obstacles by flexing or extending their knees when they encountered obstacles.

SUMMARY:
We aimed to investigate the effects of virtual reality based rehabilitation program on patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Sixty volunteer participants with knee osteoarthritis aged 40 to 65 years who were at stage of 2-3 according to the Kellgren Lawrence radiological evaluation were included in the study.

Participants were randomly divided into two groups as virtual and control group. While a conventional physiotherapy program consisting of electrotherapy and exercise program was applied to both groups 5 days a week for 6 weeks, a virtual reality program was added to the virtual group for 6 weeks, 5 days a week. At the beginning of the treatment and at the end of the sixth week, ROM, pain, kinesiophobia, proprioception, balance, muscle strength and functional status were evaluated between groups.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarhritis aged 40 to 75 years who were at stage of 2-3 according to the Kellegren Lawrence radiological evaluation were included in the study.

Exclusion Criteria:

* Those who have received physical therapy in the last 6 months
* Having serious systemic and cardiovascular diseases that may prevent exercise
* Neurological and orthopedic problems affecting gait
* Those with sensory defects
* Malignancy diagnosed
* Those who have received PRP (Platelet-Rich Plasma) treatment or intra-articular steroid injection treatment in the last 6 months
* With metal implants
* Serious hearing loss or visual impairment
* Communication problems

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Postural Balance | Change from baseline postural balance at week 6.
  PEDALO® Sensamove Balance System was used to evaluate postural balance of subjects.It has a balance board in which consists of sensors to record and process data about balance performance to a computer.
Severity of the knee Osteoarthritis | Change from baseline severity of knee osteoarthritis at week 6.
  Severity of the knee Osteoarthritis of participants was evaulated with "Western Ontario and McMaster Universities Arthritis" (WOMAC LK 3.1). The WOMAC LK has 24 questions in three subscales (pain , stiffness, physical functions) and a total of 24 questions. Each item is scored 0 to 4. Maxiumum score is 96. the higher the scores indicate that the severity of the disease is worse.
Kinesiophobia | Change from baseline kinesiophobia at week 6.
  Kinesiophobia was assessed with TAMPA Scale for Kinesiophobia (TSK). TSK is a 17-item measure that assesses kinesiophobia (fear of movement). Each item is evaluated on a 4-point Likert scale with scoring alternatives ranging from 'strongly disagree' to 'strongly agree. Total scores range from 17 to 68, with higher scores reflecting greater kinesiophobia.
Muscle Strength of Knee extensor and flexor Muscles | Change from baseline muscle strength at week 6.
  Muscle Strength was evaulated with Biodex System Pro 4 Isokinetic Dynamometer (Biodex Medical Systems, Inc, Shirley, NY. USA). The subjects were seated in such a position that knee and hip were at 900 flexion, and shoulders, ankle and pelvis were fixed to the machine. The centre of the knee joint was aligned with the centre of the dynamometer by using a laser-pointing device. Before testing, 5-min warming programme was performed by using treadmill. Isokinetic test was performed with 5 repetitions at 1200/s and 2400/s angular velocities. Tests were performed in a standardized order and all subjects have received identical instructions and encouragements.
Knee Pain | Change from baseline knee pain at week 6.
  Pain was evaulated with VAS (Visual Analog Scale). The VAS consists of a 10 cm straight line which presents a continuum of intensity and has verbal anchors at opposite ends representing 'no pain' at the bottom and 'pain as bad as it can be' at the top. The participants were asked to mark the representing point of their pain levels. The values were recorded in cm .
Knee Proprioception | Change from baseline knee proprioception at week 6.
  Knee proprioception was evaulated with MarVAJED system (Marmara Visual Auditory Joint Education Device). MarVAJED® is used in virtual rehabilitation and also has test software which can evaluate knee proprioception. The sensors of the system were placed on the upper and lower parts of the knee joint. The subjects were asked to lie down in prone position. The system was calibrated and then the knee joint was passively flexed at 30 degree. Participants were allowed to wait for ten minutes in this position to perceive the degree of knee flexion. Then the knee joint was passively brought back to the initial position and the patients were asked to actively flex their knee at 300 with their eyes closed. The same protocol was performed in 60 degree. . The difference between the reference degree and the degree that the subject performed during the test was automatically calculated by the MarVAJED system.
Range of Motion (ROM) | Change from baseline Range of Motion (ROM) at week 6.
  The active range of motion of knee (flexion, extension) was assessed by using a universal goniometer. Kendall-McCreary criteria was considered in the assessments. Measurements were repeated three times and the average value was used in the statistical analysis.
Functionality | Change baseline from functionality at week 6.
  Functionality of participants was evaulated with Aggregated Locomotor Function (ALF) test. Aggregated Locomotor Function (ALF) test consists of three parts: stair climbing, walk and transfer tests. The time was recorded for each of the tests. longer periods mean that functionality is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No